CLINICAL TRIAL: NCT00654277
Title: Comparative, Randomized, Single-Dose, Cross Over Bioavailability of Kali's Ondansetron 8 mg ODT With That of GlaxoSmithKine's Zofran 8 mg ODT in Healthy, Male and Female Subjects Under Fasting Conditions
Brief Title: Bioavailability Study of Ondansetron Orally Disintegrating Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Dr. Alfred Elvin/ Director Biopharmacetics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ODO-P2-158
Record Dates: First submitted 2008-04-03; First posted 2008-04-07 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: bioequivalence; Ondansetron ODT; Fasting; To determine bioequivalence under fasting conditions
MeSH Terms: conditions — Fasting | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received Kali formulated products under fasting conditions
  Interventions: Drug: Ondansetron
- B (Active Comparator): Subjects received GlaxoSmithKine product under fasting conditions
  Interventions: Drug: Zofran

INTERVENTIONS:
Drug: Ondansetron — ODT, 8 mg, single-dose
  Other Names: Zofran
  Arms: A
Drug: Zofran — ODT, 8 mg, fasting conditions
  Other Names: Ondansetron ODT
  Arms: B

SUMMARY:
To compare the single-dose bioavailability of Ondansetron 8 mg oDT and Zofran 8 mg ODT

DETAILED DESCRIPTION:
To Compare the single-dose bioavailability of Kali's Ondansetron 8 mg ODT with that of GlaxoSmithKine's Zofran 8 mg ODT under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following criteria may be included in the study.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form duly signed by the subject.
* Males and Females aged from 18 to 50 years ol with a body mass index (BMI)within 19-30; demographic data (sex, age, ethnic group, body weight, height and smoking habits) will be recorded and reported in the final report.
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance and must be recorded as such in the CRF (laboratory tests are presented in section 7.1.3.
* Healthy according to the laboratory results and physical examination.
* Normal cardiovascular function according to ECG.
* Non or ex-smokers.

Exclusion Criteria:

* Significant history of hypersensitivity to ondansetron or any related products as well as severe hypersensitivity reactions (like angioedema) to any drugs.
* Presence or history of significant gastrointestinal, liver or kidney disease, or any conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
* Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease.
* Females who are pregnant, lactating or are likely to become pregnant during the study phases.
* Females of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the body.
* Positive pregnancy test before and during the study.
* Maintenance therapy with any drug, or significant history or drug dependancy, alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic), or serious psychological disease.
* Any clinically significant illness in the previous 28 days before day 1 of this study.
* Use of enzyme-modifying drugs in the previous 28 days before 1 day of this study (all barbiturates, corticosteroids, phenylhydantoins, etc.).
* Participation in another clinical trial in the previous 28 days before day 1 of this study.
* Donation of 500 mL of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study.
* Positive urine screening of drugs of abuse (drug names are presented in section 7.1.4).
* Positive results to HIV, HBsAg or anti-HCV tests.
* History of fainting upon blood sampling.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2002-08; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Christian Aumais, Principal Investigator — Algotithme Pharma Inc